CLINICAL TRIAL: NCT02218593
Title: WREX Outcome Study
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Tariq Rahman, Prinicipal Research Engineer, Nemours Children's Clinic
Other Study IDs: 579772-2
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Muscular Dystrophy; Arthrogryposis; Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Dystrophies; Arthrogryposis; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WREX orthosis: When the subject used the WREX Orthosis
  Interventions: Device: WREX orthosis

INTERVENTIONS:
Device: WREX orthosis — Upper extremity exoskleton used to assist movement

SUMMARY:
This study is to evaluate how the Wilmington Robotic Exoskeleton (WREX) is working for children who are using the WREX, or have used it in the past. The survey consists of a set of questions a) performed online and b) performed over the phone.

DETAILED DESCRIPTION:
The WREX (Wilmington Robotic EXoskeleton) is being used by many children with neuromuscular conditions such as arthrogryposis and muscular dystrophy. Nemours/A.I. duPont Hospital for Children alone has provided a WREX for about 80 children in the last 3 years. This is being done through the orthopedic and muscle clinics in the hospital. We would like to perform a retrospective study to see how well the children are doing with the WREX. We propose getting this feedback through a survey administered to families using the WREX. The survey will be performed in two parts. 1) A phone survey will use the Canadian Occupational Performance Measure (COPM). 2) an online survey with additional questions. The parents are asked to submit answers on behalf of the children if they are unable to.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular disease
* Use the Wilmington Robotic Exoskeleton

Exclusion Criteria:

* people who do not use the Wilmington Robotic Exoskeleton

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People with Neuromuscular disease who use the Wilmington Robotic Exoskleton
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- WREX Orthosis: Children answering with WREX orthosis
Period: Overall Study
Arm/Group | WREX Orthosis
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- WREX Orthosis: Children who have used a WREX Orthosis
  WREX orthosis: Upper extremity exoskeleton used to assist arm movement
Arm/Group | WREX Orthosis
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.72 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Canadian Occupational Performance Measure (COPM)
Description: Performance score on The Canadian Occupational Performance Measure (COPM). The total score range is 1-10. A score of 1 indicates indicates poor performance and low satisfaction and 10 indicates good performance and high satisfaction. The numbers indicate scores on a scale.
Time Frame: Surveys were conducted at a single timepoint for each subject. The surveys were administered over a 4-month period for all the subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WREX Orthosis
Number analyzed (Participants) | 25
score on a scale | 7.09 (2.15)

ADVERSE EVENTS:
Arm/Group | WREX Orthosis
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes